CLINICAL TRIAL: NCT06160518
Title: Technology and Children's Health: Effect of Virtual Reality on Pain and Clinical Outcomes During Hydrotherapy for Children With Burn
Brief Title: Virtual Reality, Pain, Clinical Outcomes, Hydrotherapy, Children, Burn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matrouh University (Other)
Responsible Party: Principal Investigator, Seham El-Sayed Saleh Hassan, Lecturer of pediatric nursing, Matrouh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0517
Record Dates: First submitted 2023-09-20; First posted 2023-12-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Burn; Hydrotherapy
Keywords: Virtual Reality; Pain; Clinical Outcomes; Hydrotherapy; Children; Burn
MeSH Terms: conditions — Burns; Pain

STUDY DESIGN:
Intervention Model Description: virtual reality intervention which will take place using a cell phone coupled with the three-dimensional image glasses. The cell phone will play three-dimensional games which will be downloaded for free. The options for images and games involved which children could choose freely, all games will be suitable for the age group of the study.
  • The intervention will be applied for three days when hydrotherapy session done
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The children will receive the standard pharmacological treatment of the unit to manage pain and stabilize their physiological parameters throughout the three days of study.
- Study group (Experimental): The children will receive virtual reality intervention which will take place using a cell phone coupled with the three-dimensional image glasses. The cell phone will play three-dimensional games which will be downloaded for free. The options for images and games involved which children could choose freely, all games will be suitable for the age group of the study.
  Interventions: Behavioral: Virtual reality

INTERVENTIONS:
Behavioral: Virtual reality — artificial construction of 3D environment via mobile technology. It included a head-mounted device (HMD) with 3D-enabled goggles, sensory input devices and headphones, which together allow a multisensory experience to divert a child's attention.
  Arms: Study group

SUMMARY:
This study aims to evaluate the effect of virtual reality on pain and clinical outcomes during hydrotherapy for children with burn.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 3-6 years.
* Children who do not have a burned face.
* Undergoing hydrotherapy procedure for wound care.
* Able to score their own pain, with or without a visual tool.
* Willing to participate in the study.

Exclusion Criteria:

* Are cognitive or visual impairment.
* Received strong pain killer or sedative medication.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Physiological parameters assessment sheet: respiratory rate | • 10 minutes before hydrotherapy session. • 5 minutes after hydrotherapy session started without VR. • 5 minutes after hydrotherapy session started using VR. • Immediately before hydrotherapy session VR. • 10 minutes after the hydrotherapy session.
  cycle per minure
Physiological parameters assessment sheet heart rate | • 10 minutes before hydrotherapy session. • 5 minutes after hydrotherapy session started without VR. • 5 minutes after hydrotherapy session started using VR. • Immediately before hydrotherapy session VR. • 10 minutes after the hydrotherapy session.
  beat per minute
Physiological parameters assessment sheet:O2 saturation. | • 10 minutes before hydrotherapy session. • 5 minutes after hydrotherapy session started without VR. • 5 minutes after hydrotherapy session started using VR. • Immediately before hydrotherapy session VR. • 10 minutes after the hydrotherapy session.
  More than 95%
The clinical data assessment sheet:cause of burn, total body surface area burned, location of the burn, number of wounds, and the number of hydrotherapy sessions already undergoing. | • 10 minutes before hydrotherapy session. .
  clinical data

SECONDARY OUTCOMES:
Pain Assessment Scale | • 10 minutes before hydrotherapy session. • 5 minutes after hydrotherapy session started without VR. • 5 minutes after hydrotherapy session started using VR. • Immediately before hydrotherapy session VR. • 10 minutes after the hydrotherapy session.
  The behavioral/observational pain scale that adopted from (Merkel et al, 1997) will be used in this study to evaluate the children's pain intensity using the FLACC categories. Each of the five categories (F)face, (L) Legs, (A) Activity, (C) Cry, (C) Consol ability, is scored 0-2, which result in total pain rating scale 0-10 (0 = no pain, relaxed and comfortable, 10 = severe pain/discomfort).

CONTACTS AND LOCATIONS:
Locations (1):
- Matrouh university, Marsá Maţrūḩ, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali RR, Selim AO, Abdel Ghafar MA, Abdelraouf OR, Ali OI. Virtual reality as a pain distractor during physical rehabilitation in pediatric burns. Burns. 2022 Mar;48(2):303-308. doi: 10.1016/j.burns.2021.04.031. Epub 2021 May 5. PMID 34154898
- [Background] Ang SP, Montuori M, Trimba Y, Maldari N, Patel D, Chen QC. Recent Applications of Virtual Reality for the Management of Pain in Burn and Pediatric Patients. Curr Pain Headache Rep. 2021 Jan 14;25(1):4. doi: 10.1007/s11916-020-00917-0. PMID 33443603
- [Background] Centers for Disease Control and Prevention [CDC], (2019). WISQARS data visualization. Available at: https://wisqars-viz.cdc.gov:8006/lcd/home (Accessed on 1 August 2023)
- [Background] D'Alessandro, L.N., Corrales, I.L., Klein, S., Kondo, D., & Stinson, J. (2022). Using virtual reality distraction during wound management: A brief case report in a patient with epidermolysis bullosa. Pediatric Pain Letter,24(1):1-7.
- [Background] Dumoulin S, Bouchard S, Ellis J, Lavoie KL, Vezina MP, Charbonneau P, Tardif J, Hajjar A. A Randomized Controlled Trial on the Use of Virtual Reality for Needle-Related Procedures in Children and Adolescents in the Emergency Department. Games Health J. 2019 Aug;8(4):285-293. doi: 10.1089/g4h.2018.0111. Epub 2019 May 24. PMID 31135178
- [Background] Eijlers R, Utens EMWJ, Staals LM, de Nijs PFA, Berghmans JM, Wijnen RMH, Hillegers MHJ, Dierckx B, Legerstee JS. Systematic Review and Meta-analysis of Virtual Reality in Pediatrics: Effects on Pain and Anxiety. Anesth Analg. 2019 Nov;129(5):1344-1353. doi: 10.1213/ANE.0000000000004165. PMID 31136330
- [Background] Elrod J, Schiestl CM, Mohr C, Landolt MA. Incidence, severity and pattern of burns in children and adolescents: An epidemiological study among immigrant and Swiss patients in Switzerland. Burns. 2019 Aug;45(5):1231-1241. doi: 10.1016/j.burns.2019.02.009. Epub 2019 May 13. PMID 31097353
- [Background] Garrido-Ardila EM, Santos-Dominguez M, Rodriguez-Mansilla J, Torres-Piles ST, Rodriguez-Dominguez MT, Gonzalez-Sanchez B, Jimenez-Palomares M. A Systematic Review of the Effectiveness of Virtual Reality-Based Interventions on Pain and Range of Joint Movement Associated with Burn Injuries. J Pers Med. 2022 Jul 31;12(8):1269. doi: 10.3390/jpm12081269. PMID 36013218
- [Background] Gerceker GO, Bektas M, Aydinok Y, Oren H, Ellidokuz H, Olgun N. The effect of virtual reality on pain, fear, and anxiety during access of a port with huber needle in pediatric hematology-oncology patients: Randomized controlled trial. Eur J Oncol Nurs. 2021 Feb;50:101886. doi: 10.1016/j.ejon.2020.101886. Epub 2020 Dec 1. PMID 33321461
- [Background] Hansen JK, Voss J, Ganatra H, Langner T, Chalise P, Stokes S, Bhavsar D, Kovac AL. Sedation and Analgesia During Pediatric Burn Dressing Change: A Survey of American Burn Association Centers. J Burn Care Res. 2019 Apr 26;40(3):287-293. doi: 10.1093/jbcr/irz023. PMID 30844056
- [Background] Hoffman HG, Rodriguez RA, Gonzalez M, Bernardy M, Pena R, Beck W, Patterson DR, Meyer WJ 3rd. Immersive Virtual Reality as an Adjunctive Non-opioid Analgesic for Pre-dominantly Latin American Children With Large Severe Burn Wounds During Burn Wound Cleaning in the Intensive Care Unit: A Pilot Study. Front Hum Neurosci. 2019 Aug 8;13:262. doi: 10.3389/fnhum.2019.00262. eCollection 2019. PMID 31440148
- [Background] Jeschke MG, van Baar ME, Choudhry MA, Chung KK, Gibran NS, Logsetty S. Burn injury. Nat Rev Dis Primers. 2020 Feb 13;6(1):11. doi: 10.1038/s41572-020-0145-5. PMID 32054846
- [Background] Khadra C, Ballard A, Dery J, Paquin D, Fortin JS, Perreault I, Labbe DR, Hoffman HG, Bouchard S, LeMay S. Projector-based virtual reality dome environment for procedural pain and anxiety in young children with burn injuries: a pilot study. J Pain Res. 2018 Feb 14;11:343-353. doi: 10.2147/JPR.S151084. eCollection 2018. PMID 29491717
- [Background] Khadra C, Ballard A, Paquin D, Cotes-Turpin C, Hoffman HG, Perreault I, Fortin JS, Bouchard S, Theroux J, Le May S. Effects of a projector-based hybrid virtual reality on pain in young children with burn injuries during hydrotherapy sessions: A within-subject randomized crossover trial. Burns. 2020 Nov;46(7):1571-1584. doi: 10.1016/j.burns.2020.04.006. Epub 2020 May 7. PMID 32389349
- [Background] LoBiondo-Wood, G., Haber, J., & Titler, M. G. (2018). Evidence-based practice for nursing and healthcare quality improvement. Elsevier Health Sciences.
- [Background] McDonnell N. Immersive Technology and Medical Visualisation: A Users Guide. Adv Exp Med Biol. 2019;1156:123-134. doi: 10.1007/978-3-030-19385-0_9. PMID 31338782
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Norouzkhani N, Chaghian Arani R, Mehrabi H, Bagheri Toolaroud P, Ghorbani Vajargah P, Mollaei A, Hosseini SJ, Firooz M, Falakdami A, Takasi P, Feizkhah A, Saber H, Ghaffarzade H, Nemalhabib A, Ghaffari A, Osuji J, Mobayen M, Karkhah S. Effect of Virtual Reality-Based Interventions on Pain During Wound Care in Burn Patients; a Systematic Review and Meta-Analysis. Arch Acad Emerg Med. 2022 Oct 24;10(1):e84. doi: 10.22037/aaem.v10i1.1756. eCollection 2022. PMID 36426174
- [Background] Scapin S, Echevarria-Guanilo ME, Boeira Fuculo Junior PR, Goncalves N, Rocha PK, Coimbra R. Virtual Reality in the treatment of burn patients: A systematic review. Burns. 2018 Sep;44(6):1403-1416. doi: 10.1016/j.burns.2017.11.002. Epub 2018 Feb 1. PMID 29395400
- [Background] Smith KL, Wang Y, Colloca L. Impact of Virtual Reality Technology on Pain and Anxiety in Pediatric Burn Patients: A Systematic Review and Meta-Analysis. Front Virtual Real. 2022 Jan;2:751735. doi: 10.3389/frvir.2021.751735. Epub 2022 Jan 6. PMID 36247202
- [Background] Sohn D, Ring D, Toy KA, Julian JA, Arnstein P. Pain Relief and the Opioid Crisis in the United States and Canada. Instr Course Lect. 2019;68:639-646. PMID 32032104
- [Background] Won AS, Bailey J, Bailenson J, Tataru C, Yoon IA, Golianu B. Immersive Virtual Reality for Pediatric Pain. Children (Basel). 2017 Jun 23;4(7):52. doi: 10.3390/children4070052. PMID 28644422
- [Background] World Health Organization [WHO], (2018). Burns. Available at: https://www.who.int/en/news-room/fact-sheets/detail/burns (Accessed on 30 July 2023)
- [Background] Xiang H, Shen J, Wheeler KK, Patterson J, Lever K, Armstrong M, Shi J, Thakkar RK, Groner JI, Noffsinger D, Giles SA, Fabia RB. Efficacy of Smartphone Active and Passive Virtual Reality Distraction vs Standard Care on Burn Pain Among Pediatric Patients: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jun 1;4(6):e2112082. doi: 10.1001/jamanetworkopen.2021.12082. PMID 34152420